CLINICAL TRIAL: NCT00189761
Title: A Phase 2, Open-Label, Multi-Center Study to Assess Efficacy, Safety and Pharmacokinetics of a Tacrolimus New Oral Formulation (MR4) in De Novo Bone Marrow Transplant Recipients
Brief Title: A Study to Assess Efficacy, Safety and Pharmacokinetics of a Tacrolimus New Oral Formulation (MR4) in BMT Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FJ-506E-BT01
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2006-09-20 (Estimated); Status verified 2006-09

CONDITIONS: Bone Marrow Transplantation; Graft Versus Host Disease; Graft-Vs-Host Disease; Graft-Versus-Host Disease
Keywords: Tacrolimus; Immunosuppression; Bone Marrow Transplantation; Graft versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus

SUMMARY:
A study to assess efficacy, safety and pharmacokinetics of a tacrolimus new oral formulation (MR4) in de novo bone marrow transplant recipients

ELIGIBILITY:
Inclusion Criteria:

* Bone marrow transplantation patients aged 20-54 except for transplanted from genetically HLA matched sibling donor.
* The patient had been fully informed.

Exclusion Criteria:

* The patient had severe impaired hepatic function.
* The patient had impaired renal function.
* The patient had existing complication of severe cardiac dysfunction.
* The patient had severe impaired pulmonary function.

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Clinical development, Study Chair — Astellas Pharma Inc., Japan
Locations (4):
- Japan (4):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kyusyu Region